CLINICAL TRIAL: NCT00306488
Title: A Phase II Study of OT-551 Antioxidant Eye Drop in Participants With Bilateral Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: OT-551 Antioxidant Eye Drops to Treat Geographic Atrophy in Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Eye Institute (NEI) (NIH); Othera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060116; 06-EI-0116 (Other: National Eye Institute)
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2011-08

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration; AMD
Keywords: Retinal Pigment Epithelium; Dynamic Light Scattering (DLS); Visual Acuity Decrease; Intra-ocular Pressure; Autofluorescence of Retina; Age-Related Macular Degeneration; AMD
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OT-551 antioxidant eye drop (Experimental): The fellow eye was treated with OT-551 antioxidant eye drops over the course of the study.
  Interventions: Drug: OT-551 antioxidant eye drop

INTERVENTIONS:
Drug: OT-551 antioxidant eye drop — 0.45% concentration of OT-551 eye drops were given three times a day on participants with geographic atrophy area for up to three years. Participants had one eye randomized to receive the eye drop and the fellow eye was observed.

SUMMARY:
Othera Pharmaceuticals' Othera (OT)-551 antioxidant eye drop has the potential for chronic treatment of the dry form of age-related macular degeneration. This pilot study of up to 10 eye drop tolerant participants with bilateral geographic atrophy is designed to characterize the effect of 0.45% concentration of OT-551 eye drops given 3 times a day on the progression of geographic atrophy area over a two-year period. Participants will have one eye randomized to receive the eye drop and the fellow eye will be observed only.

DETAILED DESCRIPTION:
Age-related macular Degeneration (AMD), the leading cause of blindness in people over age 55 in the U.S., is a heterogeneous clinical entity in which retinal degeneration occurs predominantly in the macula in the context of aging and leads to impairment primarily of central visual acuity. AMD occurs in two general forms, one of which involves subchoroidal neovascularization with subsequent formation of a disciform scar. A second form, and the subject of this study, is termed "dry" or atrophic macular degeneration and involves a constellation of clinical features that can include drusen, pigment clumping and/or retinal pigment epithelium (RPE) dropout, and geographic atrophy. Geographic atrophy can begin as a thinning of the RPE with involvement of the underlying choriocapillaris and lead subsequently to an atrophic change in the macula. The only therapy for persons with atrophic AMD is an oral supplement containing high doses of antioxidants and zinc, which was tested by the National Eye Institute (NEI) in a large, multicenter, double-masked, placebo-controlled clinical trial with average participant follow-up of about 6 years. This antioxidant therapy was shown to modestly retard the progression of dry AMD from an intermediate stage to the advanced stages and demonstrated the benefit of antioxidant therapy in this disease.

In this study, we will evaluate Othera Pharmaceuticals' OT-551 antioxidant eye drop for chronic treatment of the dry form of AMD. This single-center, open-label, study of up to 10 participants with bilateral geographic atrophy is designed to characterize the safety of 0.45 percent concentration of OT-551 eye drops, given 3 times a day, on participants with geographic atrophy area for up to three years. Participants will have one eye randomized to receive the eye drop and the fellow eye will be observed.

ELIGIBILITY:
Inclusion Criteria

1. Participant must understand and sign the protocol's informed consent document (if the participant's vision is impaired to the point where it is not possible to read the informed consent document, the informed consent document will be read in its entirety to the participant).
2. Participant must be able to administer the eye drops or have a caretaker administer the eye drops.
3. Participant must have geographic atrophy (GA) present in both eyes compatible with age-related macular degeneration (AMD). GA is defined as one or more well-defined, usually more or less circular patches of partial or complete depigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round-ish patch of RPE partial depigmentation may still be classified as early GA. The GA in each eye must be able to be photographed in their entirety and not contiguous with any areas of peripapillary atrophy, which can complicate area measurements.
4. Participant must have a steady fixation in the study eye in the foveal or parafoveal area and media clear enough for good quality photographs.
5. Female participants of child bearing potential (those who are not post-menopausal or surgically sterile) may participate if they are not lactating and if they agree to adequate birth control methods.

4.5 Exclusion Criteria

1. Participant is > 60 years of age (to minimize fundus changes from causes other than AMD).
2. Participant is in another investigational study and actively receiving study therapy.
3. Participant is unable to comply with study procedures or follow-up visits.
4. Participant has evidence of ocular disease other than AMD in either eye that may confound the outcome of the study (e.g., diabetic retinopathy, uveitis, etc.).
5. Participant has a chronic requirement (e.g., ≥ four weeks at a time) for ocular medications for diseases, that in the judgment of the examining physician, are vision threatening or may affect the primary outcome (artificial tears are permitted).
6. Participant has evidence of pseudovitelliform macular degeneration that may confound the outcome of the study in either eye.
7. Participant with evidence of vitreo-retinal traction maculopathy that may confound the outcome of the study in either eye.
8. Participant has a history of laser, photodynamic therapy (PDT), intravitreal injection of any agent (e.g., anti-VEGF, triamcinolone, etc.), or any previous treatment for AMD other than AREDS or equivalent supplement formulation in the study eye.
9. Participant has had a vitrectomy, penetrating keratoplasty, trabeculectomy or trabeculoplasty.
10. Participant has undergone lens removal in the last three months.
11. Participant is on chemotherapy.
12. Participant is on ocular or systemic medications known to be toxic to the lens, retina, or optic nerve.
13. Participant with a history of malignancy that would compromise the 2-year study survival.
14. Participant with a history of ocular Herpes simplex virus.
15. Participant with a history of or demonstration of allergy to benzakonium chloride, a preservative agent used in the eye drop.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wai Wong, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Age-Related Eye Disease Study Research Group. A randomized, placebo-controlled, clinical trial of high-dose supplementation with vitamins C and E, beta carotene, and zinc for age-related macular degeneration and vision loss: AREDS report no. 8. Arch Ophthalmol. 2001 Oct;119(10):1417-36. doi: 10.1001/archopht.119.10.1417. PMID 11594942
- [Background] Klein R, Klein BE, Jensen SC, Meuer SM. The five-year incidence and progression of age-related maculopathy: the Beaver Dam Eye Study. Ophthalmology. 1997 Jan;104(1):7-21. doi: 10.1016/s0161-6420(97)30368-6. PMID 9022098
- [Background] Klein R, Klein BE, Linton KL. Prevalence of age-related maculopathy. The Beaver Dam Eye Study. Ophthalmology. 1992 Jun;99(6):933-43. doi: 10.1016/s0161-6420(92)31871-8. PMID 1630784
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300
- [Derived] Meleth AD, Mettu P, Agron E, Chew EY, Sadda SR, Ferris FL, Wong WT. Changes in retinal sensitivity in geographic atrophy progression as measured by microperimetry. Invest Ophthalmol Vis Sci. 2011 Feb 28;52(2):1119-26. doi: 10.1167/iovs.10-6075. Print 2011 Feb. PMID 20926818
- [Derived] Wong WT, Kam W, Cunningham D, Harrington M, Hammel K, Meyerle CB, Cukras C, Chew EY, Sadda SR, Ferris FL. Treatment of geographic atrophy by the topical administration of OT-551: results of a phase II clinical trial. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6131-9. doi: 10.1167/iovs.10-5637. Epub 2010 Jun 23. PMID 20574018

RESULTS

PARTICIPANT FLOW:
Groups:
- OT-511 Antioxidant Eye Drop: The study eye was treated with one drop (40µL) of 0.45% OT-551 antioxidant eye drops three times a day. The fellow eye was not treated with the study medication (OT-511 antioxidant eye drops).
Period: Overall Study
Arm/Group | OT-511 Antioxidant Eye Drop
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participant Information
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.91 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: The Change in Best-corrected Visual Acuity (BCVA) From Baseline to Year 2 for All Participants.
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. This acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters the Snellen measurement is 20/20.
Time Frame: 2 years
Population: Data collected from the 10 participants that completed the 24-month follow-up visit were analyzed.
  Ten study eyes and 10 fellow eyes were analyzed.
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Groups:
- Study Eye: OT-511 Antioxidant Eye Drop: The study eye was treated with one drop (40µL) of 0.45% OT-551 antioxidant eye drops three times a day.
- Fellow Eye: The fellow eye was not treated with the study medication (OT-511 antioxidant eye drops).
Arm/Group | Study Eye: OT-511 Antioxidant Eye Drop | Fellow Eye
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 10 | 10
ETDRS Letters | 0.2 (13.3) | -11.3 (7.6)

2. Secondary Outcome: The Change in Geographic Atrophy (GA), as Measured on Fundus Autofluorescence Imaging Using a Confocal Scanning Ophthalmoscope (HRA FAF) From Baseline to Year 2.
Description: Geographic Atrophy (GA), or the death of photoreceptors and surrounding cells in the retina, is a common condition in patients with Age-Related Macular Degeneration (AMD). The death of these photoreceptors results in lesions that cause vision loss. The amount of GA is measured from images produced via a non-invasive technique called Fundus Autofluorescence Imaging, which uses a Confocal Scanning Ophthalmoscope to detect the naturally-fluorescing lipofuscin (the waste that is left behind by dead photoreceptors and digested by surrounding cells) that is prevalent at the border of the lesion.
Time Frame: 2 years
Population: Data collected from the ten participants that completed the full twenty-four months of the study were analyzed.
  Ten study eyes and ten fellow eyes were analyzed.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Study Eye: OT-511 Antioxidant Eye Drop | Fellow Eye
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 10 | 10
mm^2 | 2.17 (0.83) | 2.24 (0.91)

3. Secondary Outcome: The Change in GA, as Measured on Stereoscopic Color Fundus Photography (CFP) From Baseline to Year 2.
Description: GA was also measured using Stereoscopic Color Fundus Photography (CFP), which produces color images of the inside of the eye.
Time Frame: 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Eyes
Arm/Group | Study Eye: OT-511 Antioxidant Eye Drop | Fellow Eye
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 10 | 10
mm^2 | 2.46 (1.25) | 2.47 (0.73)

4. Secondary Outcome: The Change in Contrast Sensitivity as Measured by the Pelli-Robson Chart From Baseline to Year 2.
Description: The Pelli-Robson Chart is comprised of 10 groups of 3 large letters with levels of contrast ranging from 100% (black against white) to 1% (very light gray against white). Each eye is assigned a score based on the contrast of the last group in which two or three letters were correctly read. A score of 2 log units, which represents a normal sensitivity contrast, indicates that the eye was able to detect two of the three letters with a contrast of 1 percent (contrast sensitivity = 100 percent or log 2).
Time Frame: 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log Units
Units Other Than Participants: Eyes
Arm/Group | Study Eye: OT-511 Antioxidant Eye Drop | Fellow Eye
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 10 | 10
Log Units | 0.075 (0.33) | -0.15 (0.27)

5. Secondary Outcome: Number of Participants With an Increase in the Number of Scotomatous Points Between Study and Fellow Eyes From Baseline to Year 2.
Description: Scotomatous points are testing points on microperimetry examination that are centered on the macula and report a lack of retinal sensitivity within the range tested.
Time Frame: 2 years
Population: Data were only collected in 8 of the 10 participants that completed the full 24 months. Eight study eyes and eight fellow eyes were analyzed.
Measure: Number; unit: participants
Arm/Group | Study Eye: OT-511 Antioxidant Eye Drop | Fellow Eye
Number analyzed (Participants) | 8 | 8
participants | 7 | 7

6. Secondary Outcome: The Change in Total Drusen Area From Baseline to Year 2.
Time Frame: Baseline, 2 years
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Study Eye: OT-511 Antioxidant Eye Drop | Fellow Eye
Number analyzed (Participants) | 10 | 10
mm^2 | -0.09 (0.22) | -0.06 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between December 2006 through May 2010.
Arm/Group | Participant Adverse Event Information
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participant Adverse Event Information (N=11)
Retinal haemmorhage (Eye disorders) | 4 (5)
Intraocular pressure increased (Investigations) | 1 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Mole excision (Surgical and medical procedures) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Cataract subcapsular (Eye disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Basal cell carcinoma (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Squamas cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Oedema mouth (Gastrointestinal disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Knee arthoplasty (Surgical and medical procedures) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Nerve root injury cervical (Injury, poisoning and procedural complications) | 1 (1)
Start of new cholesterol-lowering medication (Metabolism and nutrition disorders) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No